CLINICAL TRIAL: NCT03309917
Title: The Effect of Blood Pressure on Cerebral Blood Flow During Propofol Anesthesia
Acronym: CA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Niels Damkjær Olesen, Principal investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-17021598-61256
Record Dates: First submitted 2017-10-09; First posted 2017-10-16 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Gastrointestinal Neoplasms; Anesthesia, General
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Changes in mean arterial pressure (Experimental): The study is conducted from one hour after incision and lasts for approximately half an hour. Measurements are conducted at three levels of mean arterial pressure:
  * MAP set at 80-85 mmHg for 5 min.
  * MAP set at 70-75 mmHg for 5 min.
  * MAP set at 60-65 mmHg for 5 min.
  Blood pressure control is by infusion of noradrenaline. When the evaluations have been conducted blood pressure control is according to clinical practice. Measurements include internal carotid artery blood flow, mean arterial pressure, heart rate, stroke volume, frontal lobe and muscle oxygenation, depth of anesthesia, and arterial and central venous blood gas variables.
  Interventions: Other: MAP set at 80-85 mmHg for 5 min; Other: MAP set at 70-75 mmHg for 5 min; Other: MAP set at 60-65 mmHg for 5 min

INTERVENTIONS:
Other: MAP set at 80-85 mmHg for 5 min — MAP is set at 80-85 mmHg for 5 min by infusion of noradrenaline.
Other: MAP set at 70-75 mmHg for 5 min — MAP is set at 70-75 mmHg for 5 min by infusion of noradrenaline.
Other: MAP set at 60-65 mmHg for 5 min — MAP is set at 60-65 mmHg for 5 min by infusion of noradrenaline.

SUMMARY:
General anesthesia often reduces blood pressure whereby blood flow to the brain and other vital organs may become insufficient. Thus, medicine is often administered to maintain blood pressure but it is unclear at what level blood pressure should be aimed at during anesthesia.

Thirty patients undergoing major abdominal surgery will be included. The study will start one hour after the start of surgery and lasts for approximately half an hour. The purpose of the study is to evaluate whether blood flow to the brain can be increased by maintaining blood pressure at a higher level than that used in clinical practice. In the study, MAP is adjusted to a high, moderate, and low level for a short time. The low level of blood pressure used in the study, corresponds to the level aimed at in clinical practice. The drug noradrenaline will be used to control blood pressure. Blood flow to the brain will be evaluated on the neck using ultrasound.

DETAILED DESCRIPTION:
Background Propofol anesthesia reduces cerebral blood flow (CBF) and mean arterial pressure (MAP) but it is unclear whether the decrease in CBF is accentuated by hypotension. Cerebral autoregulation is generally considered to maintain CBF when MAP is between 60-150 mmHg. Hence, vasoactive medication is administered if MAP decreases to below approximately 60 mmHg.

It is controversial whether there is a plateau for cerebral autoregulation. Thus, middle cerebral artery blood velocity (MCA Vmean), as an index of CBF, is associated to MAP during pharmacological changes in MAP between approximately 40-125 mmHg. Similarly, CBF is affected by pharmacological changes in MAP between 40-80 mmHg during hypothermic cardiopulmonary bypass surgery in propofol anesthesia. Arterial hypertension may increase the lower limit of cerebral autoregulation which can be mitigated by antihypertensive treatment.

Cognitive dysfunction and delirium are common following major surgery, particularly in the elderly, and may be related to hypotension and cerebral hypoperfusion. Further, hypotensive anesthesia is associated with an increase in markers of neuronal damage, but studies have been too small to detect any difference in incidence of cognitive dysfunction following hypotensive as compared to normotensive anesthesia.

In young healthy adults, propofol anesthesia causes limited reduction in blood pressure and decreases CBF by approximately 50% by a reduction in neuronal activity. An increase in MAP from approximately 80 to 100 mmHg during propofol anesthesia does not affect CBF but it is unknown whether CBF can be increased by an increase in MAP from approximately 60 to 80 mmHg. Propofol appears to maintain cerebral autoregulation but it is unknown whether the lower level of cerebral autoregulation is affected. The internal carotid artery supplies most of CBF and dilates during moderate hypotension with maintained blood flow which indicates that the vessel contributes to cerebral autoregulation. Further, central blood volume and cardiac output may be important factors for maintaining CBF.

The study will include thirty patients planned for major abdominal surgery in propofol-remifentanil anesthesia combined with epidural analgesia. Internal carotid artery blood flow will be evaluated on the neck using duplex ultrasound. The study will be conducted one hour after the start of surgery and lasts for approximately half an hour. In the study, MAP is set pharmacologically at 80-85, 70-75 and 60-65 mmHg for a short time in random order. The level of 60-65 mmHg corresponds to the level at which MAP is maintained in clinical practice. Control of MAP is by intravenous infusion of noradrenaline, an α- and β-adrenergic agonist.

Objective The purpose of the study is to evaluate whether internal carotid artery blood flow is increased by maintaining MAP at a higher level than that used in clinical practice. Further, we evaluate whether a lower limit of cerebral autoregulation can be detected by comparing the slopes of linear regression of internal carotid artery blood flow and MAP at the evaluations when MAP is 60-65 and 70-75 mmHg and when MAP is 70-75 and 80-85 mmHg.

Hypotheses

* Internal carotid artery blood flow is higher when MAP is 80-85 mmHg as compared to a MAP of 60-65 mmHg.
* Internal carotid artery blood flow is higher when MAP is 70-75 mmHg as compared to a MAP of 60-65 mmHg.
* Internal carotid artery blood flow is higher when MAP is 80-85 mmHg as compared to a MAP of 70-75 mmHg.
* The slope of linear regression between changes in MAP and internal carotid artery blood flow is higher for the evaluations at a MAP of 70-75 and 60-65 mmHg than for the evaluations at a MAP of 80-85 and 70-75 mmHg.

Methods The study is a single-center, prospective cohort study of thirty consecutive patients planned for major abdominal surgery in propofol anesthesia. In case surgery is cancelled, or if gas anesthesia is used the patient will be excluded and excluded patients will be replaced. The number of drop-outs is expected to be between zero to five patients. Patients will be recruited the day before surgery, at which time the internal carotid artery will be evaluated using ultrasound. In case the vessel cannot be visualized, e.g. due to high localization of the carotid bifurcation the patient will not be able to participate in the study.

Anesthesia and surgery are according to clinical practice. Anesthesia is induced by propofol and maintained by propofol and remifentanil. A thoracic epidural catheter is placed at Th8/9 or Th9/10 and epidural anesthesia is initiated before surgery by bupivacaine infusion 0.5%, 5 ml/hr. and bolus 15 mg bupivacaine that is repeated hourly. Stroke volume is optimized after induction of anesthesia by repeated administration of 250 ml 5% human albumin until the increase in stroke volume is less than 10%, and volume optimization is repeated in case of persistent decrease in stroke volume by more than 10%. Noradrenaline infusion (0.6 µg/kg*ml) is started after induction of anesthesia to maintain MAP above 60 mmHg and to avoid volume optimization when the circulation is dilated.

Development of a so-called mesenteric traction syndrome can affect MAP in the first hour of major abdominal surgery. Thus, the study is conducted from 60 min after incision and lasts for approximately half an hour. Anesthesia reduces MAP, but the reduction varies between patients and is affected by administration of propofol, remifentanil, and epidural anesthesia, fluid status, and surgical stimulation etc. The start of the study is postponed until any larger bleeding, transfusion or volume optimization is treated or finished. Before the start of the study, the infusion speed of propofol and remifentanil must have been constant for at least 10 min, and at least 15 min must have elapsed since the last bolus dose bupivacaine, as any changes in anesthesia may affect both cerebral and central hemodynamics. In case the infusion of propofol or remifentanil is changed or bolus bupivacaine is administered during the study, the experiment is halted, and the study is restarted when the anesthesia has been stable for 10 min. The experiment can only be restarted once and only data from the last trial with the highest number of evaluations are used.

In the experiment MAP is temporally set to 80-85, 70-75, and 60-65 mmHg by adjusting the infusion of noradrenaline. The order of evaluations is randomized by drawing an envelope just before the start of the experiment. Noradrenaline is short lasting and have no direct effect on CBF. The experiment lasts approximately 30 min until evaluations have been conducted at the three levels of MAP. If MAP does not drop to 60-65 mmHg by halting the infusion of noradrenaline this evaluation is not conducted but we expect that this will be the case in only few patients. In clinical practice noradrenaline is used to maintain MAP > 60 mmHg. The study is not an investigation of medicinal products as noradrenaline is used as a tool to control MAP.

Administration of noradrenaline is by a central venous or large peripheral catheter, using an electronic infusion pump, and infusion speed is adjusted slowly until the level of MAP is reached. Noradrenaline is effective within 1-2 min after administration and the effect lasts only for a few minutes. When MAP has been stable at the desired level for at least 3 min, measurements are conducted during the following 2 min. When the study is finished, control of MAP will be according to clinical practice. We consider that there is no increased risk by a short term increase in MAP to 80-85 mmHg.

Measurements Arterial and central venous pressure are determined invasively while stroke volume, cardiac output, and total peripheral resistance are evaluated by modified pulse-contour analysis of the arterial pressure curve (Nexfin, BMEYE, Holland). Cerebral and biceps muscle oxygenation are evaluated using near-infrared spectroscopy (INVOS 5100C, Somanetics, Troy, MI, USA). Depth of anesthesia is assessed by Bispectral Index (BIS Complete Monitoring Systems, Covidien, USA).

Internal carotid artery blood flow is evaluated unilaterally on the neck using duplex ultrasound (Logiq E, GE Medical System, Jiangsu, Kina). Evaluation is in the longitudinal section at least 1.5 cm distal to the carotid bifurcation with the head turned approximately 30⁰ to the contralateral side. In order to limit the influence of ventilation, three recordings of approximately 15-20 s are conducted at each level of MAP and the mean is reported. A frequency of 8-12 MHz is used and gain is set as high as possible while vessel lumen is echo-free. Ultrasonic adjustments are not changed during the study. Diameter is assessed using automatic software to track the vessel wall (Brachial Analyser for Research v. 6, Medical Imaging Applications LLC, Coralville, IA, USA). The angle-corrected time maximum flow velocity (TAVMAX) is evaluated using pulsed-wave Doppler at an angle of insonation ≤ 60º. The TAVMAX corresponds to twice the mean blood velocity and blood flow is: 0.125*60*TAVMAX*π*diameter^2. Arterial and central venous blood is sampled for gas analysis and internal carotid artery blood flow is corrected for changes in PaCO2 using a factor of 3%/mmHg.

Statistics Trial size: The minimal clinically important difference in internal carotid artery blood flow between evaluations at MAP 60-65 and 80-85 mmHg is considered to be 10% as evaluations using near-infrared spectroscopy indicate that intraoperative cerebral deoxygenation of > 10% associates to postoperative cognitive function.

A power calculation indicated that at least 18 patients were required to detect a difference in internal carotid artery blood flow of 10% corresponding to 19 ml/min assuming a standard deviation for the change of 27 ml/min (unpublished results from the study "Cerebral Blood Flow During Propofol Anaesthesia" NCT02951273) to obtain a 5% significance level and a power of 80%. We plan to include 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient planned for Whipple's surgery or total pancreatic resection
* Age > 18 years

Exclusion Criteria:

* No informed consent
* Alcohol intake ≥ 420 g / week
* Beard on the neck
* Visualization of the internal carotid artery not possible, e.g. due to high placement of the bifurcation
* Stenosis that obstructs ≥ 16% of the internal carotid artery
* Cardiac disease, including congestive heart failure (NYHA II-IV), myocardial infarction, valvular heart disease or atrial fibrillation
* Neurologic disease considered to affect cerebral blood flow, including dementia, epilepsy, and apoplexy
* Intake of moclobemide, isocarboxazid or tricyclic antidepressants

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
Change in internal carotid artery blood flow when mean arterial pressure (MAP) is set to 80-85 and 60-65 mmHg | Values are recorded during 2 min at 2 time points; when MAP is set to 80-85 and 60-65 mmHg during propofol anesthesia as part of the study. The evaluations are separated by approximately 30 min
  Internal carotid artery blood flow [ml/min] assessed by duplex ultrasound when MAP is set to 80-85 and 60-65 mmHg for 5 min as part of the experiment during propofol anesthesia

SECONDARY OUTCOMES:
Change in internal carotid artery blood flow when MAP is set to 70-75 and 60-65 mmHg | Values are recorded during 2 min at 2 time points; when MAP is set to 70-75 and 60-65 mmHg during propofol anesthesia as part of the study. The evaluations are separated by approximately 15 min
  Internal carotid artery blood flow [ml/min] assessed by duplex ultrasound when MAP is set to 70-75 and 60-65 mmHg for 5 min as part of the experiment during propofol anesthesia
Change in internal carotid artery blood flow when MAP is set to 80-85 and 70-75 mmHg | Values are recorded during 2 min at 2 time points; when MAP is set to 80-85 and 70-75 mmHg during propofol anesthesia as part of the study. The evaluations are separated by approximately 15 min
  Internal carotid artery blood flow [ml/min] assessed by duplex ultrasound when MAP is set to 80-85 and 70-75 mmHg for 5 min as part of the experiment during propofol anesthesia
Comparison of the slope of linear regression of MAP and internal carotid artery blood flow for the evaluations when MAP is set to 80-85 and 70-75 mmHg and that of the evaluations when MAP is set to 70-75 and 60-65 mmHg | Values are recorded during 2 min at 3 time points; when MAP is set to 80-85, 70-75, and 60-65 mmHg during propofol anesthesia as part of the study. The evaluations are separated by approximately 15 and 30 min
  Internal carotid artery blood flow [ml/min] assessed by duplex ultrasound and MAP [mmHg] determined by radial artery cannulation when MAP is set to 80-85, 70-75, and to 60-65 mmHg for 5 min as part of the experiment during propofol anesthesia. The slope of linear regression of MAP and internal carotid artery blood flow is determined for the evaluations when MAP is set to 80-85 and 70-75 mmHg and for the evaluations when MAP is set to 70-75 and 60-65 mmHg, respectively, and the slopes are compared

CONTACTS AND LOCATIONS:
Overall Officials: Niels H Secher, MD, D.M.Sc., Study Chair — Department of Anesthesia, Rigshospitalet 2043, DK-2100 Copenhagen Ø, Denmark
Locations (1):
- Department of Anaesthesia, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi WS, Samman N. Risks and benefits of deliberate hypotension in anaesthesia: a systematic review. Int J Oral Maxillofac Surg. 2008 Aug;37(8):687-703. doi: 10.1016/j.ijom.2008.03.011. Epub 2008 Jun 3. PMID 18511238
- [Background] Ederberg S, Westerlind A, Houltz E, Svensson SE, Elam M, Ricksten SE. The effects of propofol on cerebral blood flow velocity and cerebral oxygen extraction during cardiopulmonary bypass. Anesth Analg. 1998 Jun;86(6):1201-6. doi: 10.1097/00000539-199806000-00011. PMID 9620503
- [Background] Evans DH. On the measurement of the mean velocity of blood flow over the cardiac cycle using Doppler ultrasound. Ultrasound Med Biol. 1985 Sep-Oct;11(5):735-41. doi: 10.1016/0301-5629(85)90107-3. PMID 2932831
- [Background] Greenfield JC Jr, Tindall GT. Effect of norepinephrine, epinephrine, and angiotensin on blood flow in the internal carotid artery of man. J Clin Invest. 1968 Jul;47(7):1672-84. doi: 10.1172/JCI105858. PMID 4298077
- [Background] Kaisti KK, Metsahonkala L, Teras M, Oikonen V, Aalto S, Jaaskelainen S, Hinkka S, Scheinin H. Effects of surgical levels of propofol and sevoflurane anesthesia on cerebral blood flow in healthy subjects studied with positron emission tomography. Anesthesiology. 2002 Jun;96(6):1358-70. doi: 10.1097/00000542-200206000-00015. PMID 12170048
- [Background] KETY SS, KING BD, HORVATH SM, JEFFERS WS, HAFKENSCHIEL JH. The effects of an acute reduction in blood pressure by means of differential spinal sympathetic block on the cerebral circulation of hypertensive patients. J Clin Invest. 1950 Apr;29(4):402-7. doi: 10.1172/JCI102272. No abstract available. PMID 15415440
- [Background] Kristensen SD, Knuuti J, Saraste A, Anker S, Botker HE, Hert SD, Ford I, Gonzalez-Juanatey JR, Gorenek B, Heyndrickx GR, Hoeft A, Huber K, Iung B, Kjeldsen KP, Longrois D, Luscher TF, Pierard L, Pocock S, Price S, Roffi M, Sirnes PA, Sousa-Uva M, Voudris V, Funck-Brentano C; Authors/Task Force Members. 2014 ESC/ESA Guidelines on non-cardiac surgery: cardiovascular assessment and management: The Joint Task Force on non-cardiac surgery: cardiovascular assessment and management of the European Society of Cardiology (ESC) and the European Society of Anaesthesiology (ESA). Eur Heart J. 2014 Sep 14;35(35):2383-431. doi: 10.1093/eurheartj/ehu282. Epub 2014 Aug 1. No abstract available. PMID 25086026
- [Background] LASSEN NA. Cerebral blood flow and oxygen consumption in man. Physiol Rev. 1959 Apr;39(2):183-238. doi: 10.1152/physrev.1959.39.2.183. No abstract available. PMID 13645234
- [Background] Li S, Hoskins PR, Anderson T, McDicken WN. Measurement of mean velocity during pulsatile flow using time-averaged maximum frequency of Doppler ultrasound waveforms. Ultrasound Med Biol. 1993;19(2):105-13. doi: 10.1016/0301-5629(93)90002-6. PMID 8516956
- [Background] Lucas SJ, Tzeng YC, Galvin SD, Thomas KN, Ogoh S, Ainslie PN. Influence of changes in blood pressure on cerebral perfusion and oxygenation. Hypertension. 2010 Mar;55(3):698-705. doi: 10.1161/HYPERTENSIONAHA.109.146290. Epub 2010 Jan 18. PMID 20083726
- [Background] Matta BF, Lam AM, Strebel S, Mayberg TS. Cerebral pressure autoregulation and carbon dioxide reactivity during propofol-induced EEG suppression. Br J Anaesth. 1995 Feb;74(2):159-63. doi: 10.1093/bja/74.2.159. PMID 7696064
- [Background] Meng L, Hou W, Chui J, Han R, Gelb AW. Cardiac Output and Cerebral Blood Flow: The Integrated Regulation of Brain Perfusion in Adult Humans. Anesthesiology. 2015 Nov;123(5):1198-208. doi: 10.1097/ALN.0000000000000872. PMID 26402848
- [Background] Newman MF, Croughwell ND, Blumenthal JA, White WD, Lewis JB, Smith LR, Frasco P, Towner EA, Schell RM, Hurwitz BJ, et al. Effect of aging on cerebral autoregulation during cardiopulmonary bypass. Association with postoperative cognitive dysfunction. Circulation. 1994 Nov;90(5 Pt 2):II243-9. PMID 7955260
- [Background] Olesen J. The effect of intracarotid epinephrine, norepinephrine, and angiotensin on the regional cerebral blood flow in man. Neurology. 1972 Sep;22(9):978-87. doi: 10.1212/wnl.22.9.978. No abstract available. PMID 4343348
- [Background] Olesen J. Beta-adrenergic effects on cerebral circulation. Cephalalgia. 1986;6 Suppl 5:41-6. doi: 10.1177/03331024860060S505. PMID 2879631
- [Background] Olesen J, Paulson OB, Lassen NA. Regional cerebral blood flow in man determined by the initial slope of the clearance of intra-arterially injected 133Xe. Stroke. 1971 Nov-Dec;2(6):519-40. doi: 10.1161/01.str.2.6.519. No abstract available. PMID 5164581
- [Background] Olesen ND, Sorensen H, Ambrus R, Svendsen LB, Lund A, Secher NH. A mesenteric traction syndrome affects near-infrared spectroscopy evaluated cerebral oxygenation because skin blood flow increases. J Clin Monit Comput. 2018 Apr;32(2):261-268. doi: 10.1007/s10877-017-0014-2. Epub 2017 Mar 14. PMID 28293809
- [Background] Panerai RB. Assessment of cerebral pressure autoregulation in humans--a review of measurement methods. Physiol Meas. 1998 Aug;19(3):305-38. doi: 10.1088/0967-3334/19/3/001. PMID 9735883
- [Background] Patti R, Saitta M, Cusumano G, Termine G, Di Vita G. Risk factors for postoperative delirium after colorectal surgery for carcinoma. Eur J Oncol Nurs. 2011 Dec;15(5):519-23. doi: 10.1016/j.ejon.2011.01.004. Epub 2011 Feb 17. PMID 21333597
- [Background] Siepe M, Pfeiffer T, Gieringer A, Zemann S, Benk C, Schlensak C, Beyersdorf F. Increased systemic perfusion pressure during cardiopulmonary bypass is associated with less early postoperative cognitive dysfunction and delirium. Eur J Cardiothorac Surg. 2011 Jul;40(1):200-7. doi: 10.1016/j.ejcts.2010.11.024. Epub 2010 Dec 18. PMID 21168339
- [Background] Song XX, Yu BW. Anesthetic effects of propofol in the healthy human brain: functional imaging evidence. J Anesth. 2015 Apr;29(2):279-88. doi: 10.1007/s00540-014-1889-4. Epub 2014 Jul 24. PMID 25056258
- [Background] Strandgaard S. Autoregulation of cerebral blood flow in hypertensive patients. The modifying influence of prolonged antihypertensive treatment on the tolerance to acute, drug-induced hypotension. Circulation. 1976 Apr;53(4):720-7. doi: 10.1161/01.cir.53.4.720. PMID 815061
- [Background] Strebel S, Lam AM, Matta B, Mayberg TS, Aaslid R, Newell DW. Dynamic and static cerebral autoregulation during isoflurane, desflurane, and propofol anesthesia. Anesthesiology. 1995 Jul;83(1):66-76. doi: 10.1097/00000542-199507000-00008. PMID 7605020
- [Background] Strebel SP, Kindler C, Bissonnette B, Tschaler G, Deanovic D. The impact of systemic vasoconstrictors on the cerebral circulation of anesthetized patients. Anesthesiology. 1998 Jul;89(1):67-72. doi: 10.1097/00000542-199807000-00012. PMID 9667295
- [Background] Thomas KN, Lewis NC, Hill BG, Ainslie PN. Technical recommendations for the use of carotid duplex ultrasound for the assessment of extracranial blood flow. Am J Physiol Regul Integr Comp Physiol. 2015 Oct;309(7):R707-20. doi: 10.1152/ajpregu.00211.2015. Epub 2015 Jul 8. PMID 26157060
- [Background] Willie CK, Macleod DB, Shaw AD, Smith KJ, Tzeng YC, Eves ND, Ikeda K, Graham J, Lewis NC, Day TA, Ainslie PN. Regional brain blood flow in man during acute changes in arterial blood gases. J Physiol. 2012 Jul 15;590(14):3261-75. doi: 10.1113/jphysiol.2012.228551. Epub 2012 Apr 10. PMID 22495584
- [Background] Lin R, Zhang F, Xue Q, Yu B. Accuracy of regional cerebral oxygen saturation in predicting postoperative cognitive dysfunction after total hip arthroplasty: regional cerebral oxygen saturation predicts POCD. J Arthroplasty. 2013 Mar;28(3):494-7. doi: 10.1016/j.arth.2012.06.041. Epub 2012 Nov 12. PMID 23151365
- [Background] Mille T, Tachimiri ME, Klersy C, Ticozzelli G, Bellinzona G, Blangetti I, Pirrelli S, Lovotti M, Odero A. Near infrared spectroscopy monitoring during carotid endarterectomy: which threshold value is critical? Eur J Vasc Endovasc Surg. 2004 Jun;27(6):646-50. doi: 10.1016/j.ejvs.2004.02.012. PMID 15121117
- [Background] Jiang X, Chen D, Lou Y, Li Z. Risk factors for postoperative delirium after spine surgery in middle- and old-aged patients. Aging Clin Exp Res. 2017 Oct;29(5):1039-1044. doi: 10.1007/s40520-016-0640-4. Epub 2016 Oct 20. PMID 27766513
- [Background] Lin S, McKenna SJ, Yao CF, Chen YR, Chen C. Effects of Hypotensive Anesthesia on Reducing Intraoperative Blood Loss, Duration of Operation, and Quality of Surgical Field During Orthognathic Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Oral Maxillofac Surg. 2017 Jan;75(1):73-86. doi: 10.1016/j.joms.2016.07.012. Epub 2016 Jul 25. PMID 27542543
- [Background] Liu J, Zhu YS, Hill C, Armstrong K, Tarumi T, Hodics T, Hynan LS, Zhang R. Cerebral autoregulation of blood velocity and volumetric flow during steady-state changes in arterial pressure. Hypertension. 2013 Nov;62(5):973-9. doi: 10.1161/HYPERTENSIONAHA.113.01867. Epub 2013 Sep 16. PMID 24041946
- [Background] Newman S, Stygall J, Hirani S, Shaefi S, Maze M. Postoperative cognitive dysfunction after noncardiac surgery: a systematic review. Anesthesiology. 2007 Mar;106(3):572-90. doi: 10.1097/00000542-200703000-00023. PMID 17325517
- [Derived] Olesen ND, Frederiksen HJ, Storkholm JH, Hansen CP, Svendsen LB, Olsen NV, Secher NH. Internal carotid artery blood flow is enhanced by elevating blood pressure during combined propofol-remifentanil and thoracic epidural anaesthesia: A randomised cross-over trial. Eur J Anaesthesiol. 2020 Jun;37(6):482-490. doi: 10.1097/EJA.0000000000001189. PMID 32175988

DOCUMENTS (2):
  • Study Protocol (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT03309917/Prot_002.pdf
  • Statistical Analysis Plan (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT03309917/SAP_003.pdf